CLINICAL TRIAL: NCT00108069
Title: A Phase II Trial of Tamoxifen and Bortezomib in Patients With Recurrent High-Grade Gliomas
Brief Title: Tamoxifen and Bortezomib to Treat Recurrent Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine E. Warren, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 050137; 05-C-0137; NCT00112762 (obsolete NCT alias)
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Glioma
Keywords: Brain; Tumor; Malignant; Therapy; Progression; Chemotherapy; Antiangiogenesis; Radiation; Malignant Brain Tumor; Malignant Glioma; Glioma
MeSH Terms: conditions — Glioma; Neoplasms; Disease Progression; Brain Neoplasms | interventions — Tamoxifen; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBM (Glioblastoma multiforme) (Experimental)
  Interventions: Drug: Tamoxifen citrate; Drug: Bortezomib
- AG (Anaplastic glioma) (Experimental)
  Interventions: Drug: Tamoxifen citrate; Drug: Bortezomib

INTERVENTIONS:
Drug: Tamoxifen citrate — oral dose 120 mg twice a day, every day
  Other Names: Nolvadex
Drug: Bortezomib — intravenous (IV) injection 1.3 mg/m^2 days 3, 6, 10, 13, 24, 27,31,34 on every 6 week cycle
  Other Names: Velcade

SUMMARY:
This study will determine whether the drugs tamoxifen and bortezomib can delay tumor growth in patients with recurrent glioma (malignant brain tumor). Tamoxifen may work by interfering with the internal signaling needed for the cancer to grow. Bortezomib may also interfere with tumor growth processes. Laboratory studies show that low doses of bortezomib significantly enhance glioma cell death when used with tamoxifen.

Patients 18 years of age and older with glioma whose tumor does not respond to standard medical treatment and who are not taking enzyme-inducing anti-seizure medications such as Dilantin, phenobarbitol, or Tegretol, may be eligible for this study. Candidates are screened with a physical examination, blood tests, and magnetic resonance imaging (MRI) or computed tomography (CT). MRI and CT scans produce images of the brain that can show if the brain tumor is growing (see below).

Participants receive treatment in 6-week cycles for up to 1 year. (The treatment duration may be extended in some patients who continue to tolerate the drug and show no signs of tumor growth after 1 year.) During each cycle, patients take six tamoxifen tablets twice a day every day and receive bortezomib by infusion into a vein on days 3, 6, 10, 13, 24, 27, 31 and 34. Treatment may continue as long as the tumor does not grow and the patient does not develop unacceptable side effects. In addition to drug treatment, patients undergo the following tests and procedures:

* Periodic routine blood tests.
* MRI or CT scan of the head before starting each new cycle. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. CT uses x-rays to provide 3-dimensional views of the part of the body being studied. For both procedures, the patient lies on a table that slides into the cylindrical scanner.
* Blood test to measure levels of bortezomib. Blood is drawn before the bortezomib infusion on days 3 and 24, and 4 hours after the infusion on day 24 of the first treatment cycle only.
* Dynamic MRI with spectroscopy or positron emission tomography (PET). Patients may be asked to undergo one of these tests, which help distinguish live tumor from dying tumor. The experience of dynamic MRI with spectroscopy is the same as standard MRI and is done at the same time as the standard procedure (see above). PET uses a radioactive substance to show cellular activity in specific tissues of the body. The patient is given an injection of a sugar solution in which a radioactive isotope has been attached to the sugar molecule. A special camera detects the radiation emitted by the radioisotope, and the resulting images show how much glucose is being used in various parts of the body. Because rapidly growing cells, such as tumors, take up and use more glucose than normal cells do, this test can be used to show active tumors.
* Drug diary. Patients maintain a calendar to record when they take their study drugs and what side effects they develop.

DETAILED DESCRIPTION:
Background:

Tamoxifen (TAM), a member of the selective estrogen receptor modulator (SERM) family, is widely used in the treatment of estrogen receptor (ER) expressing breast cancer. It has previously been shown that high-dose TAM has cytotoxic activity against glioma cells, but whether this effect is drug-specific or represents a general property of SERMs was unknown. We have now demonstrated that suppression of nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) activation markedly enhances SERM-induced apoptosis, suggesting a role for NF-kB in protecting glioma cells from SERM-induced cytotoxicity.

Bortezomib is a potent inhibitor of the 26S proteosome and causes significant anti-proliferative and cytotoxic effects in a number of cell lines through its protean effects on a variety of cellular signaling pathways, including its ability to potently inhibit the NF-kB pathway. We have recently demonstrated that bortezomib has significant anti-glioma activity in vitro and a ongoing clinical trial has demonstrated some possible activity in patients with recurrent gliomas. We have now also generated preclinical data demonstrating that bortezomib in combination with Tamoxifen has synergistic cytotoxic effects on glioma cells.

Thus, given the minimal to modest activity of both drugs in patients with recurrent gliomas, given their spectrum of non-overlapping toxicities, and given the marked synergistic glioma cell killing of the combination of drugs in our preclinical screens, we are now proposing a phase II trial of bortezomib in combination with Tamoxifen in patients with recurrent gliomas not taking enzyme inducing anti-epileptic drugs (EIAEDs).

Objectives:

The primary statistical endpoint will be response (defined as either stable disease or objective response as is standard in neuro-oncology clinical trials) after 6 weeks of treatment.

Eligibility:

Patients with histologically proven high-grade gliomas or patients with a clinical and radiographic diagnosis of brainstem glioma will be eligible for this protocol.

Design:

The phase II study will be stratified by the type of high grade glioma (anaplastic glioma (AA) or glioblastoma (GBM)) and a two-stage min-max design with a maximum of 41 patients in the GBM stratum and 36 patients in the AA stratum.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically proven high-grade gliomas or patients with a clinical and radiographic diagnosis of brainstem glioma will be eligible for this protocol. High-grade gliomas include glioblastoma multiforme (GBM; stratum 1) and its variants such as gliosarcoma and anaplastic gliomas (AG; stratum 2), such as anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma/glioma NOS (not otherwise specified).

Patients must have unequivocal evidence for tumor progression by magnetic resonance imaging (MRI) or computerized tomography (CT) scan. This scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

1. They have recovered from the effects of surgery.
2. Residual disease following resection of recurrent tumor is mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:

   * no later than 96 hours in the immediate post-operative period or
   * at least 4 weeks post-operatively, and
   * within 14 days of registration, and
   * on a steroid dosage that has been stable for at least 5 days.

   If the 96 hour scan is more than 21 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.

   Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.

   Ability of subjects or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

   Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.

   Patients must have a Karnofsky performance status of greater than or equal to 60.

   Patients must have recovered from the toxic effects of prior therapy: 2 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.

   Patients must have adequate bone marrow function (white blood cell (WBC) greater than or equal to 3,000/microl, absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, platelet count of greater than or equal to 100,000/mm^3, and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (serum glutamic oxaloacetic transaminase (SGOT) and bilirubin less than 2 times ULN), and adequate renal function (creatinine less than 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

   Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy.

   This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

   Patients must practice adequate contraception.

   EXCLUSION CRITERIA:

   Patients who, in the view of the treating physician, have significant active cardiac (documented coronary artery disease, congestive heart failure, arrhythmia requiring medication), hepatic (hepatocellular and/or cholestatic dysfunction as documented by liver biopsy, liver ultrasound, or abnormal liver function blood tests, renal (as documented by renal biopsy, ultrasound, CT/MRI scans or reflected in the blood tests or psychiatric diseases (requiring hospitalization or is of significant severity to impair the patients ability to cooperate with the study instructions).

   No concurrent use of other standard chemotherapeutics or investigative agents.

   Patients known to have an active malignancy other than their glioma (except non-melanoma skin cancer or carcinoma in-situ of the cervix).

   Patients who have an active infection requiring intravenous (IV) antibiotics.

   Patients who are pregnant or breast feeding.

   Patients who have any disease that will obscure toxicity or dangerously alter drug metabolism.

   Patients who have had clear tumor progression while being treated with tamoxifen and/or patients treated with tamoxifen within the past year.

   Patients who are taking EIAEDs (enzyme inducing anti-epileptic drugs) are not eligible.

   Patients who have had documented tumor progression while taking tamoxifen and/or any treatment with tamoxifen within 6 months of registration.

   Salicylates ARE permitted.

   Patients with grade 2 or greater peripheral neuropathy.

   Invasive procedures defined as follows:
   * Major surgical procedures, open biopsy or significant traumatic injury within 28 days prior to Day ! therapy
   * Anticipation of need for major surgical procedures during the course of the study
   * Core biopsy within 7 days prior to D1 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker D, Wright E, Nguyen K, Cannon L, Fain P, Goldgar D, Bishop DT, Carey J, Baty B, Kivlin J, et al. Gene for von Recklinghausen neurofibromatosis is in the pericentromeric region of chromosome 17. Science. 1987 May 29;236(4805):1100-2. doi: 10.1126/science.3107130.
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991
- [Derived] Odia Y, Kreisl TN, Aregawi D, Innis EK, Fine HA. A phase II trial of tamoxifen and bortezomib in patients with recurrent malignant gliomas. J Neurooncol. 2015 Oct;125(1):191-5. doi: 10.1007/s11060-015-1894-y. Epub 2015 Aug 19. PMID 26285768
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0137.html

RESULTS

PARTICIPANT FLOW:
Groups:
- GBM (Glioblastoma Multiforme); AG (Anaplastic Glioma): Bortezomib : intravenous (IV) injection 1.3 mg/m^2 days 3, 6, 10, 13, 24, 27,31,34 on every 6 week cycle
  Tamoxifen citrate : oral dose 120 mg twice a day, every day
Period: Overall Study
Arm/Group | GBM (Glioblastoma Multiforme) | AG (Anaplastic Glioma)
Started | 30 | 13
Completed | 0 | 0
Not Completed | 30 | 13
Not completed — Never rec'd study drug | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Not completed — Progessive disease | 27 | 11

BASELINE CHARACTERISTICS:
Population: One participant in the AG cohort was not evaluable/did not receive study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | GBM (Glioblastoma Multiforme) | AG (Anaplastic Glioma) | Total
Number analyzed (Participants) | 30 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 12 | 41
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 42 (10) | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 23 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 11 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 10 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Response, Defined as Stable Disease or Objective (Partial or Complete) Response.
Description: Complete response (CR) is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. All measurable, evaluable and non-evaluable lesions and site must be assessed using the same techniques as baseline. Patients who respond must be on the same or decreasing doses of dexamethasone. Partial response (PR) is greater than or equal to a 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable disease. No new lesions. All measurable and evaluable lesions and sites must be assessed using same techniques as baseline. Responders must be on the same decreasing doses of dexamethasone. Stable disease (SD) does not qualify for CR, PR, or progression (e.g., a 25% increase in the sum of products of all measurable lesions). The designation of stable/no response requires a minimum of 6 weeks duration. All measurable and evaluable sites must be assessed using the same techniques as baseline.
Time Frame: Patients were followed for an average of six weeks for assessment of response
Population: Two patients were not able to complete follow-up neuroimaging to assess response due to clinical progression of disease.
Measure: Number; unit: Participants
Arm/Group | GBM (Glioblastoma Multiforme) | AG (Anaplastic Glioma)
Number analyzed (Participants) | 28 | 12
Participants
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 1 | 0
  Progressive disease | 27 | 12

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 7.5 years
Measure: Number; unit: Participants
Arm/Group | GBM (Glioblastoma Multiforme) | AG (Anaplastic Glioma)
Number analyzed (Participants) | 30 | 12
Participants | 30 | 12

3. Secondary Outcome: Adverse Event Grades
Description: The combined serious and non-serious adverse event Table describes count of patients whose highest grade adverse event for any CTC (common terminology criteria) term was related to study drugs for the GBM (Glioblastoma multiforme) and AG (Anaplastic glioma) cohorts.
Time Frame: 7.5 years
Population: Neither cohort completed planned accrual and are small in number separately. Additionally, the underlying histological grade would not affect toxicity. Therefore, these cohorts may be combined. The Table describes count of patients whose highest grade adverse event for any CTC (common terminology criteria) term was related to study drugs.
Measure: Number; unit: participants
Groups:
- Grade 1: Mild adverse event
- Grade 2: Moderate adverse event
- Grade 3: Severe adverse event
- Grade 4: Life-threatening or disabling adverse event
- Grade 5: Death related to adverse event
- Total: Total number of participants.
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Total
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
participants
  thrombocytopenia | 19 | 3 | 1 | 1 | 0 | 24
  lymphopenia | 4 | 4 | 4 | 0 | 0 | 12
  hypophosphatemia | 0 | 6 | 3 | 0 | 0 | 9
  ALT/sGPT | 6 | 1 | 0 | 0 | 0 | 7
  anemia (Decreased Hgb) | 6 | 0 | 0 | 0 | 0 | 6
  hyponatremia | 4 | 0 | 1 | 0 | 0 | 5
  headache | 0 | 2 | 1 | 0 | 0 | 3
  leukopenia | 1 | 2 | 0 | 0 | 0 | 3
  AST/sGOT | 2 | 0 | 0 | 0 | 0 | 2
  dyspnea | 1 | 0 | 1 | 0 | 0 | 2
  fatigue | 2 | 0 | 0 | 0 | 0 | 2
  fever | 1 | 1 | 0 | 0 | 0 | 2
  hyperkalemia | 2 | 0 | 0 | 0 | 0 | 2
  cough | 1 | 0 | 0 | 0 | 0 | 1
  depression (mood alteration) | 0 | 1 | 0 | 0 | 0 | 1
  diarrhea | 0 | 1 | 0 | 0 | 0 | 1
  dizziness | 1 | 0 | 0 | 0 | 0 | 1
  venous thrombosis | 0 | 0 | 1 | 0 | 0 | 1
  edema | 1 | 0 | 0 | 0 | 0 | 1
  hyperbilirubinemia | 1 | 0 | 0 | 0 | 0 | 1
  hypermagnesemia | 1 | 0 | 0 | 0 | 0 | 1
  hypocalcemia | 1 | 0 | 0 | 0 | 0 | 1
  hypokalemia | 1 | 0 | 0 | 0 | 0 | 1
  hypotension | 1 | 0 | 0 | 0 | 0 | 1
  elevated creatinine | 1 | 0 | 0 | 0 | 0 | 1
  infection with unknown ANC | 0 | 0 | 1 | 0 | 0 | 1
  neutropenia | 0 | 1 | 0 | 0 | 0 | 1
  pain | 0 | 1 | 0 | 0 | 0 | 1
  rash | 1 | 0 | 0 | 0 | 0 | 1
  hemorrhage (rectal) | 1 | 0 | 0 | 0 | 0 | 1
  somnolence | 0 | 0 | 1 | 0 | 0 | 1
  urinary frequency | 1 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | GBM (Glioblastoma Multiforme) | AG (Anaplastic Glioma)
Serious Adverse Events (participants affected / at risk) | 11/30 | 3/12
Other Adverse Events (participants affected / at risk) | 26/30 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBM (Glioblastoma Multiforme) (N=30) | AG (Anaplastic Glioma) (N=12)
Death not associated with CTCAE term: Death NOS (General disorders) | 1 (1) | 1 (1)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 4 (4) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0)
Infection - Other (Specify, infection w/unknown ANC) (Infections and infestations) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0)
Pain: head/headache (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 1 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (2) | 1 (1)
Speech impairment (e.g., dysphagia or aphasia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vascular - Other (Specify-deep vein thrombosis) (Vascular disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC<1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1)
Muscle weakness, genralized or specific area (not due to neuropathy): Right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) — Other, specify - shingles R T9 & T10 dermatomes both anteriorly & posteriorly, w/herpetic neuralgia pain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBM (Glioblastoma Multiforme) (N=30) | AG (Anaplastic Glioma) (N=12)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Blood/Bone Marrow - Other (Specify, elevated white blood count;) (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Patient's platelets kept dropping and was 27 on 12/12, RBC-3.45, Hgb-10.6, Hct 30.8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Extremity - lower (gait-walking) (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC<1.0 x 10e9/L) (General disorders) | 1 (1) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Hypotension (Cardiac disorders) | 1 (2) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Lymphatics - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — displayed signs of bilateral edema in his feet/ankle area, lt pitting edema
Lymphopenia (Blood and lymphatic system disorders) | 10 (14) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration: depression (Nervous system disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Facial (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Right-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy): Whole-body/generalized (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 3 (5) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (2) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nystagmus (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Specify, horizontal diplopia) (Eye disorders) | 1 (1) | 0 (0)
Pain - Other (Specify, L side - hip and rib) (General disorders) | 1 (1) | 0 (0)
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain: head/headache (Nervous system disorders) | 3 (4) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (6) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 13 (21) | 4 (5)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (5) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Speech impairment (e.g., dysphagia or aphasia) (Nervous system disorders) | 7 (7) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Constitutional symptoms - Other (Specify, fatigue) (General disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemorrhage: GI: Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L): lung (pneumonia)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No